CLINICAL TRIAL: NCT01535001
Title: Structured Non-operative Treatment of Knee Osteoarthritis - a Randomized Controlled Trial of Pain, Physical Function and Quality of Life With 12months Follow-up
Brief Title: Structured Non-operative Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: The Danish Rheumatism Association (Other); Association of Danish Physiotherapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20110085
Record Dates: First submitted 2012-02-09; First posted 2012-02-17 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis, Knee; Treatment Outcome; Time Factors; Rehabilitation; Combined Modality Therapy; Middle Aged; Aged; Aged, 80 and over; Male; Female; Humans; Analysis of Variance
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acetaminophen; Pantoprazole; Nutrition Assessment; Patient Education as Topic; Foot Orthoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDIC (Active Comparator): Medicine, Exercise, Diet, Insole and Cognitive/patient education (MEDIC) for three months.
  Interventions: Other: Neuromuscular training (NEMEX-TJR); Drug: Paracetamol; Drug: Burana; Drug: Pantoprazole; Behavioral: Dietary counseling; Behavioral: Patient education; Other: Insoles
- Standard treatment (Active Comparator): Information on knee osteoarthritis, and on what they can do to treat the disorder and prevent it from being worse.
  Interventions: Behavioral: Information

INTERVENTIONS:
Other: Neuromuscular training (NEMEX-TJR) — 60min. of neuromuscular training two times a week for 3 months (12 weeks) using the neuromuscular training program called NEMEX-TJR.
  Other Names: No other
  Arms: MEDIC
Behavioral: Information — Information on knee osteoarthritis, and on what they can do to treat the disorder and prevent it from being worse.
  Information will be given in a leaflet.
  Other Names: No other
  Arms: Standard treatment
Drug: Paracetamol — 1 g x 4/day
  Other Names: No other
  Arms: MEDIC
Drug: Burana — 400 mg x 3/day for three weeks
  Other Names: No other
  Arms: MEDIC
Drug: Pantoprazole — 20mg x 1/day for three weeks
  Other Names: No other
  Arms: MEDIC
Behavioral: Dietary counseling — For participants with a BMI equal to or >25. The dietitian initiates a 3-month intervention that provides instruction and guidance in relation to diet and plans the number of visits according to the individual participant needs.
  Other Names: No other
  Arms: MEDIC
Behavioral: Patient education — The aim is to strengthen the participant's involvement in the treatment, so the participant will be in a position to handle, master and act reasonable in relation to their knee OA. This aspect of the intervention is based on principles from The Chronic Disease Self-Management Program, "Lær at leve med kronisk sygdom (Learn to live with chronic illness)" by The National Board of Health, Denmark and "Artrosskolan Spenshult" in Sweden.
  Other Names: No other
  Arms: MEDIC
Other: Insoles — The position of the knee is assessed using Single Leg Mini Squat. On the basis of this test it is decided which of two types of insoles (Formthotics System) the participant should have (neutral with a lateral wedge or neutral).
  The participants will be advised to use the insoles in all shoes.
  Other Names: No other
  Arms: MEDIC

SUMMARY:
The purpose of this study is to test whether an algorithm for systematic non-surgical treatment consisting of corrective insoles, neuromuscular training, weight loss, patient education and pharmacological treatment with paracetamol, non steroidal anti inflammatory drugs (NSAIDs) and Pantoprazole provides further improvement in pain, function and quality of life than standard non-surgical treatment (information on the disease and how to treat it) in patients with knee osteoarthritis.

The H1-hypothesis is that the treatment algorithm results in a greater increase in quality of life and functional capacity and greater reduction in pain than standard treatment at the primary endpoint, which is follow-up 12months after the start of the treatment.

See statistical analysis plan available under "Links" for further description of the study.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is the degenerative joint disease that most often requires treatment and at the same time the one associated with the greatest social costs. In addition, the disease has many personal costs and is greatly contributing to reduced functionality and autonomy of older adults.

It is recommended both nationally and internationally that the treatment of knee osteoarthritis should include multiple treatment modalities. Clinical guidelines recommend that exercise, weight loss and patient education is the first step in treatment and that insoles and pharmacological treatment can be included as a supplement.

However if the patient is not a candidate for total knee replacement, the patient most often receives only information on knee osteoarthritis, and on what they can do to treat the disorder and prevent it from being worse. This postponement of treatment can lead to a worsening of pain and function and a worse outcome after treatment. Therefore, the current treatment strategy for the patient group is problematic.

The current practice may be due to the lack of studies with high level of evidence that have examined the optimal non-operative treatment approach and compared it with the current standard treatment for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Knee-OA detected by x-ray (Kellgren & Lawrence grade 1 or greater)
* KOOS4 of ≤ 75
* Considered not to be a candidate for Total Knee Replacement (TKR) by the orthopedic surgeon.
* The participant is > 18 years of age.
* The participant can provide relevant and adequate, informed consent.

Exclusion Criteria:

* Prior TKA ipsilateral
* Rheumatoid arthritis
* Mean VAS > 60mm the last week on a 0-100mm scale
* Possible pregnancy or planning pregnancy;
* Inability to comply with the protocol;
* Inadequacy in written and spoken Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren T. Skou, PhD-student, Principal Investigator — Orthopaedic Research Unit, Aalborg University Hospital, Denmark; Ewa M. Roos, PhD, Study Chair — Research Unit for Musculoskeletal Function and Physiotherapy, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark, Denmark; Lars Arendt-Nielsen, Dr.Sci.Med., Study Chair — Center for Sensory-Motor Interaction (SMI), Department of Health Sciences and Technology, Aalborg University; Mogens B. Laursen, PhD, Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Sten Rasmussen, M.D., Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Michael S. Rathleff, PhD-student, Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Ole H. Simonsen, Dr.Sci.Med., Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark
Locations (3):
- Denmark (3):
  - Department of Occupational and Physiotherapy, Aalborg Hospital-Aarhus University Hospital, Aalborg
  - Farsoe Hospital, Farsø
  - Vendsyssel Hospital, Frederikshavn, Frederikshavn

REFERENCES:
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Fortin PR, Penrod JR, Clarke AE, St-Pierre Y, Joseph L, Belisle P, Liang MH, Ferland D, Phillips CB, Mahomed N, Tanzer M, Sledge C, Fossel AH, Katz JN. Timing of total joint replacement affects clinical outcomes among patients with osteoarthritis of the hip or knee. Arthritis Rheum. 2002 Dec;46(12):3327-30. doi: 10.1002/art.10631. PMID 12483739
- [Background] Rossi MD, Eberle T, Roche M, Waggoner M, Blake R, Burwell B, Baxter A. Delaying knee replacement and implications on early postoperative outcomes: a pilot study. Orthopedics. 2009 Dec;32(12):885. doi: 10.3928/01477447-20091020-06. PMID 19968215
- [Background] National Board of Health, Denmark. Referenceprogram for knæartrose. Copenhagen: National Board of Health, Denmark; 2007. [22.02.2010] found at: http://www.sst.dk/publ/Publ2007/PLAN/SfR/Refprg_knaeartrose.pdf
- [Background] Skou ST, Rasmussen S, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Roos EM. The efficacy of 12 weeks non-surgical treatment for patients not eligible for total knee replacement: a randomized controlled trial with 1-year follow-up. Osteoarthritis Cartilage. 2015 Sep;23(9):1465-75. doi: 10.1016/j.joca.2015.04.021. Epub 2015 Apr 30. PMID 25937024
- [Derived] Larsen JB, Roos EM, Laursen M, Holden S, Johansen MN, Rathleff MS, Arendt-Nielsen L, Rasmussen S, Skou ST. Five-year follow-up of patients with knee osteoarthritis not eligible for total knee replacement: results from a randomised trial. BMJ Open. 2022 Nov 25;12(11):e060169. doi: 10.1136/bmjopen-2021-060169. PMID 36428014
- [Derived] Skou ST, Roos EM, Laursen M, Arendt-Nielsen L, Rasmussen S, Simonsen O, Ibsen R, Larsen AT, Kjellberg J. Cost-effectiveness of 12 weeks of supervised treatment compared to written advice in patients with knee osteoarthritis: a secondary analysis of the 2-year outcome from a randomized trial. Osteoarthritis Cartilage. 2020 Jul;28(7):907-916. doi: 10.1016/j.joca.2020.03.009. Epub 2020 Mar 31. PMID 32243994
- [Derived] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Rasmussen S, Simonsen O. Total knee replacement and non-surgical treatment of knee osteoarthritis: 2-year outcome from two parallel randomized controlled trials. Osteoarthritis Cartilage. 2018 Sep;26(9):1170-1180. doi: 10.1016/j.joca.2018.04.014. Epub 2018 May 1. PMID 29723634
- [Derived] Arendt-Nielsen L, Simonsen O, Laursen MB, Roos EM, Rathleff MS, Rasmussen S, Skou ST. Pain and sensitization after total knee replacement or nonsurgical treatment in patients with knee osteoarthritis: Identifying potential predictors of outcome at 12 months. Eur J Pain. 2018 Jul;22(6):1088-1102. doi: 10.1002/ejp.1193. Epub 2018 Feb 15. PMID 29369450
- [Derived] Skou ST, Rasmussen S, Simonsen O, Roos EM. Knee Confidence as It Relates to Self-reported and Objective Correlates of Knee Osteoarthritis: A Cross-sectional Study of 220 Patients. J Orthop Sports Phys Ther. 2015 Oct;45(10):765-71. doi: 10.2519/jospt.2015.5864. Epub 2015 Aug 24. PMID 26304646
- [Derived] Skou ST, Roos EM, Simonsen O, Laursen MB, Rathleff MS, Arendt-Nielsen L, Rasmussen S. The efficacy of non-surgical treatment on pain and sensitization in patients with knee osteoarthritis: a pre-defined ancillary analysis from a randomized controlled trial. Osteoarthritis Cartilage. 2016 Jan;24(1):108-16. doi: 10.1016/j.joca.2015.07.013. Epub 2015 Aug 1. PMID 26241775
- [Derived] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. Efficacy of multimodal, systematic non-surgical treatment of knee osteoarthritis for patients not eligible for a total knee replacement: a study protocol of a randomised controlled trial. BMJ Open. 2012 Nov 14;2(6):e002168. doi: 10.1136/bmjopen-2012-002168. Print 2012. PMID 23151395
- See also: Link to the published statistical analysis plan — http://vbn.aau.dk/da/publications/statistical-analysis-plan-sap-for-medic2(3e75f67a-4333-439a-bb0b-b8e21bc19fb1).html

RESULTS

PARTICIPANT FLOW:
Groups:
- MEDIC: 60min. of neuromuscular training two times a week for 3 months (12 weeks) using the neuromuscular training program called NEMEX-TJR.
  Paracetamol: 1 g x 4/day
  Burana: 400 mg x 3/day
  Pantoprazole: 20mg x 1/day
  Dietary counseling: For participants with a BMI equal to or >25. The dietitian initiates a 3-month intervention that provides instruction and guidance in relation to diet
  Patient education: The aim is to strengthen the participant's involvement in the treatment, so the participant will be in a position to handle, master and act reasonable in relation to their knee OA.
  Insoles: The position of the knee is assessed using Single Leg Mini Squat. On the basis of this test it is decided which of two types of insoles (Formthotics System) the participant should have (neutral with a lateral wedge or neutral).
  The participants will be advised to use the insoles in all shoes.
- Standard Treatment: Information on knee osteoarthritis, and on what they can do to treat the disorder and prevent it from being worse.
  Information: Information on knee osteoarthritis, and on what they can do to treat the disorder and prevent it from being worse.
  Information will be given in a leaflet.
Period: Overall Study
Arm/Group | MEDIC | Standard Treatment
Started | 50 | 50
Completed | 47 | 44
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- MEDIC: 60min. of neuromuscular training two times a week for 3 months (12 weeks) using the neuromuscular training program called NEMEX-TJR.
  Paracetamol: 1 g x 4/day
  Burana: 400 mg x 3/day
  Pantoprazole: 20mg x 1/day
  Dietary counseling: For participants with a BMI equal to or >25. The dietitian initiates a 3-month intervention that provides instruction and guidance in relation to diet.
  Patient education: The aim is to strengthen the participant's involvement in the treatment, so the participant will be in a position to handle, master and act reasonable in relation to their knee OA.
  Insoles: The position of the knee is assessed using Single Leg Mini Squat. On the basis of this test it is decided which of two types of insoles (Formthotics System) the participant should have (neutral with a lateral wedge or neutral).
  The participants will be advised to use the insoles in all shoes.
- Total: Total of all reporting groups
Arm/Group | MEDIC | Standard Treatment | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.7) | 67.1 (9.1) | 66.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 24 | 25 | 49
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (5.6) | 29.4 (5.2) | 30.0 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in KOOS4 (Knee Injury and Osteoarthritis Outcome Score)
Description: The average score for four of the five KOOS subscales, covering pain, symptoms, difficulties in functions of daily living, and quality of life (KOOS4), with scores ranging from 0 (worst) to 100 (best).
  Between group comparisons of treatment effect (change in KOOS4 from baseline to 1 year follow-up) will be dependent on data distribution. We expect the change to be normally distributed and analysis will be made using a mixed model ANOVA with subject being a random factor and visit (baseline, 3, 6 and 12 months), treatment arm (TKA + MEDIC, MEDIC) and site (Frederikshavn, Farsoe) being fixed factors. Baseline KOOS4 will be a covariate. Furthermore interactions between the fixed factors will be included in the model. P-values and 95% CI will be presented to assess superiority.
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 50 | 50
units on a scale | 18.2 [13.0 to 23.4] | 7.1 [1.4 to 12.9]

2. Secondary Outcome: Change From Baseline in EQ-5D
Description: Between groups comparisons of the change from baseline to the 1 year follow-up in all secondary endpoint will be handled similar to the primary endpoint. See statistical analysis plan for further description (available under "Links").
  Range of EQ-5D Descriptive Index is -0.59 to 1.00 (worst to best), while the EQ VAS goes from 0 to 100 (worst to best).
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 50 | 50
units on a scale
  Descriptive index | 0.140 [0.095 to 0.186] | 0.075 [0.018 to 0.132]
  EQ VAS | 5.3 [-0.4 to 11.0] | 7.2 [0.1 to 14.2]

3. Secondary Outcome: Change From Baseline in 20-meter Walk
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: sec
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 50 | 50
sec | -1.2 [-1.6 to -0.8] | -0.6 [-1.1 to -0.1]

4. Secondary Outcome: Change in the Five KOOS Subscale Scores From Baseline
Description: Range of all subscales are 0 to 100 (worst to best).
Time Frame: Primary: 12 months.
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 50 | 50
units on a scale
  Pain | 18.7 [12.9 to 24.6] | 9.3 [2.9 to 15.6]
  Symptoms | 16.3 [10.6 to 22.0] | 7.7 [1.5 to 13.9]
  Activities of Daily Living | 18.7 [12.6 to 24.8] | 5.9 [-0.8 to 12.6]
  Sports and recreation | 16.0 [7.8 to 24.1] | 12.0 [4.8 to 19.3]
  Quality of Life | 19.0 [12.9 to 25.2] | 5.5 [-1.1 to 12.1]

5. Secondary Outcome: Weight Change in kg From Baseline
Description: Weight change in kg measured without shoes at the same time of day and on the same scale
Time Frame: Primary: 12months.
Population: Only patients with a BMI equal to or >25 were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 42 | 37
kg | -2.4 [-3.8 to -1.1] | -2.4 [-4.1 to -0.6]

6. Secondary Outcome: Proportion of Users of Pain Medication
Description: With possible answers being yes and no
Time Frame: Baseline and 12months.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 50 | 50
proportion of participants
  Baseline | 0.64 [0.50 to 0.76] | 0.56 [0.42 to 0.69]
  12months | 0.39 [0.26 to 0.54] | 0.57 [0.42 to 0.71]

7. Secondary Outcome: Number of Serious Adverse Events Reported at Index Knee
Description: Adverse events (AE) and seriously adverse events (SAE) will be registered in three ways and divided into index knee or sites other than index knee. The project physiotherapist will record any adverse events that the participant experiences or tells them about. For the participants allocated to, or crossing over to, TKA, a project worker will look through hospital records to register if any pre-defined perioperative and postoperative adverse events occurred. At all follow-ups, the assessor will use open-probe questioning to assess adverse events in all participants.
Time Frame: Primary: 12months.
Measure: Number; unit: Serious adverse events related to knee
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 50 | 50
Serious adverse events related to knee | 13 | 24

8. Secondary Outcome: Change From Baseline in Time From the Timed Up and Go
Time Frame: Primary: 12 months.
Measure: Mean (95% Confidence Interval); unit: sec
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 50 | 50
sec | -1.4 [-1.9 to -0.9] | -1.1 [-1.7 to -0.5]

9. Other Pre Specified Outcome: Exploratory Outcomes
Description: 1. Pain intensities on a 100 mm VAS with terminal descriptors of 'no pain' and 'worst pain possible' in various situations.
  2. Number of sites with pain in the previous 24 hours shaded on a region-divided body chart
  3. Pain location and type assessed using the Knee Pain Map.
  4. Maximum isometric muscle strength measured bilaterally in knee flexion and knee extension in a make test using a handheld dynamometer (Powertrack II TM Commander).
  5. Pressure pain thresholds measured bilaterally using a handheld algometer (Algometer Type II) at five sites at the knee and the m. tibialis anterior muscle and the m. extensor carpi radialis longus.
  6. Postural balance assessed using an instrumented force platform (Good Balance), measuring the centre of pressure excursion.
  7. Self-efficacy in improving pain, function and QOL in various situations using a 100 mm VAS with terminal descriptors of 'very unsure' and 'very sure'.
Time Frame: Baseline, 3months, 6months, 12months and 24months
Population: Since this is exploratory outcomes they will be analyzed in future publications.
Arm/Group | MEDIC | Standard Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | MEDIC | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 11/50 | 14/50
Other Adverse Events (participants affected / at risk) | 17/50 | 14/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC (N=50) | Standard Treatment (N=50)
Total knee replacement (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Arthrodesis of contralateral foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Erysipelas (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intestinal cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Knee arthroscopy (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Blood transfusion during TKR surgery (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
pain without loosening of the prosthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Fracture of os sacrum (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Low back pain radiating to leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Frature of collum femoris (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
heart problems (Vascular disorders) | 0 (0) | 1 (1)
severe physical decline due to influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
renal-artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Atherosclerosis demanding angioplasty (Vascular disorders) | 0 (0) | 1 (1)
canalolithiasis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Instability after TKR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Swelling after TKR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC (N=50) | Standard Treatment (N=50)
Pain in index knee (Musculoskeletal and connective tissue disorders) | 14 (14) | 12 (12)
Swelling in index knee (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Decreased range of motion in index knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Calor around index knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rubor (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Achilles Tendinopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Broken toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
foot painof short duration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
intermittent hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
sciatic nerve pain of short duration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ankle sprain (grade I) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain in the contralateral knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hamstring strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No